CLINICAL TRIAL: NCT02372344
Title: A Phase I, Single Centre, Randomized, Open-Label, Three-Period Crossover Study to Investigate the Effect of Food on Pharmacokinetics of Total EPA and Total DHA With a Single 4 g Dose of AZD0585 in Healthy Male Japanese Subjects
Brief Title: A Study to Investigate the Effect of Food on Pharmacokinetics of Total EPA and Total DHA of AZD0585 in Healthy Male Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D5884C00004
Record Dates: First submitted 2015-02-05; First posted 2015-02-26 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: the effect of food timing on PK; the effect of food timing on Safety and Tolerability; AZD0585; Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fasting (Experimental): Each subject will receive a single oral dose of 4 g AZD0585 on Day 1 of Visits 2, 3, and 4. Each dose will be administered at the end of a 10-hour fast.
  Interventions: Drug: AZD0585
- Before meal (Experimental): Each subject will receive a single oral dose of 4 g AZD0585 on Day 1 of Visits 2, 3, and 4. Each dose will be administered before consumption of a low calorie, low-fat breakfast (within 30 minutes before starting food intake).
  Interventions: Drug: AZD0585
- After meal (Experimental): Each subject will receive a single oral dose of 4 g AZD0585 on Day 1 of Visits 2, 3, and 4. Each dose will be administered after consumption of a low calorie, low-fat breakfast (within 30 minutes after starting food intake).
  Interventions: Drug: AZD0585

INTERVENTIONS:
Drug: AZD0585 — Following an overnight fast of at least 10 hours, a single dose of 4 g AZD0585 will be administered on 3 separate occasions (fasting, before meal, and after meal) in a randomized crossover fashion with different food restrictions.

SUMMARY:
The purpose of this study is to assess the effect of food timing on pharmacokinetics (PK) of AZD0585 and the effect of food timing on tolerability and safety of AZD0585 in healthy male Japanese subjects.

DETAILED DESCRIPTION:
This study is an open-label, randomized, cross-over design with three single-dose treatment periods and a washout of at least 10 days in between each treatment visit. The study period consists of 5 visits to the study centre: Visit 1 (enrolment), Visit 2 (first single-dose treatment), Visit 3 (second single-dose treatment), Visit 4 (third single-dose treatment) and Visit 5 (follow-up).

Target subject population is healthy male Japanese subjects aged 20-45 years. Following an overnight fast of at least 10 hours, a single dose of 4 g AZD0585 will be administered on 3 separate occasions (fasting, before meal, and after meal) in a randomized crossover fashion with different food restrictions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese male, 20 to 45 years of age (inclusive).
* Body mass index (BMI) ≥ 18.5 and ≤ 25 (kg/m2).
* Medically healthy with clinically insignificant screening results (e.g., laboratory profiles, medical histories, ECGs, physical findings). Hemoglobin level must be ≥ the lower limit of study centre reference range. 12-Lead ECG with QT interval corrected for heart rate using Fridericia's formula (QTcF) should be > 340 msec and < 450 msec.
* No habitual use of drug(s) and tobacco/nicotine-containing products for a minimum of 3 months prior to first dosing.
* Subjects must be willing and able to give written informed consent by signing an Institutional Review Board (IRB)-approved Informed Consent Form prior to admission to this study and follow the restrictions and procedures outlined for the study.

Exclusion Criteria:

* Past history of psychological or physical disorder which may affect the objectives of this study, in the opinion of the PI.
* An individual who has abnormal laboratory values (ie, suggesting hepatic, renal, cardiovascular or endocrine disorders or diabetes mellitus), or an inappropriate current or past medical history for participation based on the decision of the PI.
* A history or presence of significant cardiovascular, pulmonary, hepatic, renal, haematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease.
* Had used fish oil, other EPA- and/or DHA-containing supplements within 2 months prior to first admission day.
* Have serum (or plasma) EPA and/or DHA concentrations exceeding the upper limit of reference range for the "fatty acids profile, four-fraction" test, determined at Visit 1.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kei Sakamoto, MD, PhD, Principal Investigator — Sugioka Memorial Hospital, Medical Co. LTA; Torbjörn Lundström, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Fukuoka, Japan

REFERENCES:
- [Derived] Shimada H, Nilsson C, Noda Y, Kim H, Lundstrom T, Yajima T. Effects of Food on the Pharmacokinetics of Omega-3-Carboxylic Acids in Healthy Japanese Male Subjects: A Phase I, Randomized, Open-label, Three-period, Crossover Trial. J Atheroscler Thromb. 2017 Sep 1;24(9):980-987. doi: 10.5551/jat.38737. Epub 2017 Mar 24. PMID 28344197

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period started 4 March 2015 and the last subject last visit was 12 May 2015. This was a 3-period crossover study with a minimum 10-day washout period between each treatment visit (Period 1=Visit 2; Period 2=Visit 3; Period 3=Visit 4).
Pre-assignment Details: Subjects were randomized to 3 sequences (ABC, BCA or CAB; A=fasting, B=before meal, C=after meal) with a 1:1:1 ratio. 72 subjects were enrolled; 42 randomized and 30 excluded (8 did not fulfil eligibility criteria and 22 refused participation).
Groups:
- Sequence ABC: Subjects randomized to treatment sequence ABC: A=fasting / B=before meal / C=after meal.
  Following an overnight fast of at least 10 hours, a single oral dose of 4 g AZD0585 was administered on 3 separate occasions (fasting, before meal, and after meal) in a randomized crossover fashion with different food restrictions.
- Sequence BCA: Subjects randomized to treatment sequence BCA: B=before meal / C=after meal / A=fasting.
  Following an overnight fast of at least 10 hours, a single oral dose of 4 g AZD0585 was administered on 3 separate occasions (fasting, before meal, and after meal) in a randomized crossover fashion with different food restrictions.
- Sequence CAB: Subjects randomized to treatment sequence CAB: C=after meal / A=fasting / B=before meal.
  Following an overnight fast of at least 10 hours, a single oral dose of 4 g AZD0585 was administered on 3 separate occasions (fasting, before meal, and after meal) in a randomized crossover fashion with different food restrictions.
Period: Period 1 (Visit 2)
Arm/Group | Sequence ABC | Sequence BCA | Sequence CAB
Started | 14 | 14 | 14
Completed | 14 | 14 | 14
Not Completed | 0 | 0 | 0
Period: Period 2 (Visit 3)
Arm/Group | Sequence ABC | Sequence BCA | Sequence CAB
Started | 14 | 14 | 14
Completed | 14 | 14 | 14
Not Completed | 0 | 0 | 0
Period: Period 3 (Visit 4)
Arm/Group | Sequence ABC | Sequence BCA | Sequence CAB
Started | 14 | 14 | 14
Completed | 14 | 14 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects (n = 42) were included in the baseline analysis.
Groups:
- AZD0585: All subjects received a single oral dose of 4 g AZD0585 on 3 separate occasions (fasting, before meal, and after meal) in a randomized crossover fashion with different food restrictions. Each dose was administered on Day 1 of each separate treatment period: Period 1=Visit 2; Period 2=Visit 3; Period 3=Visit 4.
Arm/Group | AZD0585
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 42
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Food Timing (Fasting, Before Meal, and After Meal) on Pharmacokinetics (PK; AUC) of AZD0585 in Healthy Male Japanese.
Description: To investigate the effect of food timing on PK (area under the plasma concentration-time curve from time zero to infinity [AUC]) of single dose of 4 g AZD0585 in healthy male Japanese by assessing plasma concentrations of total eicosapentaenoic acid (EPA) and total docosahexaenoic acid (DHA), and PK parameters over time under the three proposed conditions (fasting, before meal, and after meal).
Time Frame: Blood samples were collected from pre-dose (Day -1) up to 72 hours post-dose for each of the separate treatment periods (Visits 2, 3 and 4).
Population: The PK set included all healthy subjects in the safety population (ie, who received at least 1 administration of AZD0585 and for whom any post-dose data were available) with at least 1 detectable total EPA and total DHA plasma concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram x hour /millilitre (mg⋅h/mL)
Groups:
- Fasting: Each subject received a single oral dose of 4 g AZD0585 on Day 1 of Visits 2, 3, and 4. Each dose was administered at the end of a 10-hour fast.
- Before Meal: Each subject received a single oral dose of 4 g AZD0585 on Day 1 of Visits 2, 3, and 4. Each dose was administered before consumption of a low calorie, low-fat breakfast (within 30 minutes before starting food intake).
- After Meal: Each subject received a single oral dose of 4 g AZD0585 on Day 1 of Visits 2, 3, and 4. Each dose was administered after consumption of a low calorie, low-fat breakfast (within 30 minutes after starting food intake).
Arm/Group | Fasting | Before Meal | After Meal
Number analyzed (Participants) | 37 | 33 | 41
milligram x hour /millilitre (mg⋅h/mL)
  Total EPA (n=37, 33, 41) | 2.44 (66.8) | 2.66 (80.15) | 3.80 (37.55)
  Total DHA (n=4, 2, 2) | 0.299 (143) | 0.444 (152) | 0.617 (97.7)
Statistical Analysis 1: Comparison: Fasting vs After Meal; Total EPA: Ratio of Fasting to After meal. Primary comparisons for total EPA were based on a linear mixed-effect model. This model included log-transformed PK parameter (AUC) as a response variable and treatment, sequence and period as fixed categorical effects, and subject nested within sequence as a random categorical effect; Test type: Superiority or Other; Geometric least square (LS) mean ratio = 0.64, 95% CI 2-sided [0.54 to 0.77]
Statistical Analysis 2: Comparison: Before Meal vs After Meal; Total EPA: Ratio of Before meal to After meal. Primary comparisons for total EPA were based on a linear mixed-effect model. This model included log-transformed PK parameter (AUC) as a response variable and treatment, sequence and period as fixed categorical effects, and subject nested within sequence as a random categorical effect; Test type: Superiority or Other; Geometric LS mean ratio = 0.71, 95% CI 2-sided [0.59 to 0.86]

2. Primary Outcome: The Effect of Food Timing (Fasting, Before Meal, and After Meal) on PK (Cmax) of AZD0585 in Healthy Male Japanese.
Description: To investigate the effect of food timing on PK (maximum plasma concentration [Cmax]) of single dose of 4 g AZD0585 in healthy male Japanese by assessing plasma concentrations of total EPA and total DHA, and PK parameters over time under the three proposed conditions (fasting, before meal, and after meal). Analyses of the outcome measures presented are for baseline-adjusted data for total EPA and DHA since the presence of endogenous levels of these fatty acids would likely contribute to intra-subject variability and affect the analyses and interpretation. The geometric mean was calculated as the exponential of the arithmetic mean calculated from data on a log scale.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/millilitre (mcg/mL)
Arm/Group | Fasting | Before Meal | After Meal
Number analyzed (Participants) | 42 | 42 | 42
microgram/millilitre (mcg/mL)
  Total EPA (n=42, 42, 42) | 78.5 (110) [10.9 to 271] | 97.1 (168) [6.40 to 386] | 221 (34.7) [72.2 to 378]
  Total DHA (n=42, 42, 42) | 42.1 (84.9) [11.8 to 157] | 52.4 (103) [9.73 to 178] | 92.6 (42.65) [27.0 to 195]
Statistical Analysis 1: Comparison: Fasting vs After Meal; Total EPA: Ratio of Fasting to After meal. Primary comparisons for total EPA were based on a linear mixed-effect model. This model included log-transformed PK parameter (Cmax) as a response variable and treatment, sequence and period as fixed categorical effects, and subject nested within sequence as a random categorical effect; Test type: Superiority or Other; Geometric LS mean ratio = 0.35, 95% CI 2-sided [0.27 to 0.47]
Statistical Analysis 2: Comparison: Before Meal vs After Meal; Total EPA: Ratio of Before meal to After meal. Primary comparisons for total EPA were based on a linear mixed-effect model. This model included log-transformed PK parameter (Cmax) as a response variable and treatment, sequence and period as fixed categorical effects, and subject nested within sequence as a random categorical effect; Test type: Superiority or Other; Geometric LS mean ratio = 0.44, 95% CI 2-sided [0.33 to 0.59]
Statistical Analysis 3: Comparison: Fasting vs After Meal; Total DHA: Ratio of Fasting to After meal. Primary comparisons for total DHA were based on a linear mixed-effect model. This model included log-transformed PK parameter (Cmax) as a response variable and treatment, sequence and period as fixed categorical effects, and subject nested within sequence as a random categorical effect; Test type: Superiority or Other; Geometric LS mean ratio = 0.46, 95% CI 2-sided [0.36 to 0.57]
Statistical Analysis 4: Comparison: Before Meal vs After Meal; Total DHA: Ratio of Before meal to After meal. Primary comparisons for total DHA were based on a linear mixed-effect model. This model included log-transformed PK parameter (Cmax) as a response variable and treatment, sequence and period as fixed categorical effects, and subject nested within sequence as a random categorical effect; Test type: Superiority or Other; Geometric LS mean ratio = 0.57, 95% CI 2-sided [0.45 to 0.71]

3. Primary Outcome: The Effect of Food Timing (Fasting, Before Meal, and After Meal) on PK (AUC0-72) of AZD0585 in Healthy Male Japanese.
Description: To investigate the effect of food timing on PK (area under the plasma concentration-time curve from time zero to 72 hours [AUC0-72]) of single dose of 4 g AZD0585 in healthy male Japanese by assessing plasma concentrations of total EPA and total DHA, and PK parameters over time under the three proposed conditions (fasting, before meal, and after meal). Analyses of the outcome measures presented are for baseline-adjusted data for total EPA and DHA since the presence of endogenous levels of these fatty acids would likely contribute to intra-subject variability and affect the analyses and interpretation. The geometric mean was calculated as the exponential of the arithmetic mean calculated from data on a log scale.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg⋅h/mL
Arm/Group | Fasting | Before Meal | After Meal
Number analyzed (Participants) | 42 | 42 | 42
mg⋅h/mL
  Total EPA (n=42, 42, 42) | 1.53 (76.1) [0.353 to 4.37] | 1.52 (112) [0.0682 to 4.95] | 2.76 (31.1) [0.912 to 5.04]
  Total DHA (n=42, 42, 42) | 0.542 (80.4) [0.118 to 1.55] | 0.533 (66.0) [0.111 to 1.80] | 0.621 (75.8) [0.107 to 1.86]
Statistical Analysis 1: Comparison: Fasting vs After Meal; Total EPA: Ratio of Fasting to After meal. Primary comparisons for total EPA were based on a linear mixed-effect model. This model included log-transformed PK parameter (AUC0-72) as a response variable and treatment, sequence and period as fixed categorical effects, and subject nested within sequence as a random categorical effect; Test type: Superiority or Other; Geometric LS mean ratio = 0.56, 95% CI 2-sided [0.45 to 0.69]
Statistical Analysis 2: Comparison: Before Meal vs After Meal; Total EPA: Ratio of Before Meal to After meal. Primary comparisons for total EPA were based on a linear mixed-effect model. This model included log-transformed PK parameter (AUC0-72) as a response variable and treatment, sequence and period as fixed categorical effects, and subject nested within sequence as a random categorical effect; Test type: Superiority or Other; Geometric LS mean ratio = 0.55, 95% CI [0.44 to 0.69]
Statistical Analysis 3: Comparison: Fasting vs After Meal; Total DHA: Ratio of Fasting to After meal. Primary comparisons for total DHA were based on a linear mixed-effect model. This model included log-transformed PK parameter (AUC0-72) as a response variable and treatment, sequence and period as fixed categorical effects, and subject nested within sequence as a random categorical effect; Test type: Superiority or Other; Geometric LS mean ratio = 0.87, 95% CI 2-sided [0.73 to 1.04]
Statistical Analysis 4: Comparison: Before Meal vs After Meal; Total DHA: Ratio of Before meal to After meal. Primary comparisons for total DHA were based on a linear mixed-effect model. This model included log-transformed PK parameter (AUC0-72) as a response variable and treatment, sequence and period as fixed categorical effects, and subject nested within sequence as a random categorical effect; Test type: Superiority or Other; Geometric LS mean ratio = 0.86, 95% CI 2-sided [0.72 to 1.02]

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were collected from randomisation (Visit 2, Day 1) until the follow up visit (Visit 5).
Description: Visits 2, 3 and 4 comprised 3 separate treatment periods with a washout period of at least 10 days between each treatment visit.
Arm/Group | Fasting | Before Meal | After Meal
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 5/42 | 6/42 | 1/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fasting (N=42) | Before Meal (N=42) | After Meal (N=42)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 6 (6) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Statistical analysis is not provided for the treatment comparisons of AUC for the parameter total DHA (not possible to calculate in majority of subjects). Therefore, AUC(0-72) alone represents total plasma exposure in the bioavailability comparison.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less